CLINICAL TRIAL: NCT04595058
Title: Multicenter, Randomized and Comparative Study of Lumen-apposing Metal Stents With or Without Coaxial Plastic Stent for Endoscopic Ultrasound-guided Transmural Biliary Drainage
Brief Title: LAMS Choledochoduodenostomies: With or Without Coaxial Plastic Stent
Acronym: BAMPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Hospital del Rio Hortega (Other); Hospital Clínico Universitario de Valencia (Other); Hospital General Universitario de Alicante (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Provincial de Castellon (Other)
Responsible Party: Principal Investigator, Joan B Gornals, Head of Interventional Digestive Endoscopy Unit., Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAMPI
Record Dates: First submitted 2020-09-22; First posted 2020-10-20 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2022-12

CONDITIONS: Biliary Obstruction; Pancreatic Cancer; Biliary Tract Neoplasms
Keywords: Choledochoduodenostomy;; Therapeutic endoscopy; lumen apposing metal stent; biliary drainage
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EUSDB-LAMS (Active Comparator): Endoscopic ultrasound-guided choledochoduodenostomy with lumen-apposing metal stent . Formal indication on biliopancreatic drainage according to the instruction forms of the manufacturer.
  EUSDB-LAMS (Endoscopic ultrasound guided biliary drainage with lumen-apposing metal stent)
  Interventions: Device: Lumen-apposing metal stent without double pigtail plastic stent
- EUSDB-LAMS-Pigtail (Experimental): Endoscopic ultrasound-guided choledochoduodenostomy with lumen-apposing metal stents without coaxial plastic stent. Formal indication on biliopancreatic drainage according to the instruction forms of the manufacturer.
  In this arm, a double pigtail through the lumen apposing metal stent will be inserted as an axis-orienting stent.
  EUSDB-LAMS-Pigtial (Endoscopic ultrasound guided biliary drainage with lumen-apposing metal stent (LAMS) and axis-orienting double-pigtail plastic stent through LAMS)
  Interventions: Device: Double pigtail plastic stent through lumen-apposing metal stent

INTERVENTIONS:
Device: Double pigtail plastic stent through lumen-apposing metal stent — Biliary drainage guided by endoscopic ultrasound: Addition or not, of a axis-orienting plastic stent, mostly, double-pigtail stent through the lumen of a lumen-apposing metal stent
  Arms: EUSDB-LAMS-Pigtail
Device: Lumen-apposing metal stent without double pigtail plastic stent — Endoscopic ultrasound-guided transmural biliary drainage is with lumen-apposing metal stent is a formal indication according to the instruction forms of the manufacturer.
  Arms: EUSDB-LAMS

SUMMARY:
The aim of the study is to evaluate technical, clinical and safety outcomes of lumen-apposing metal stent (LAMS) with and without a coaxial double-pigtail plastic stent (DPS) in EUS-guided choledochoduodenostomies (CDS) for the management of biliary obstruction.

DETAILED DESCRIPTION:
The introduction of specific biliary lumen-apposing metal stents (LAMS) represented a great technical improvement in EUS-guided transmural Biliary drainage (BD) of distal malignant biliary obstruction Data is still limited, but recent studies and reviews have been reported with acceptable technical and clinical success. However, some concerns exist regarding its safety, as secondary adverse events

There are doubts concerning the possible benefits derived from the insertion of double-pigtail plastic stents (DPS) within the lumen-apposing metal stents (LAMS) in the EUS-guided choledochoduodenostomy (CDS). Our hypothesis is that adding a coaxial plastic stent may offer benefits in terms of safety in CDS.

ELIGIBILITY:
Inclusion Criteria:

* Distal biliary strictures,
* A prior failed attempt at biliary drainage
* informed consent provided by the patient.

Patient exclusion criteria were as follows:

* younger than age 18 years,
* coagulopathy (international normalized ratio >1.5, marked thrombocytopenia with a platelet count <50,000/mL, or patient on anticoagulation therapy),
* critical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
Safety (Adverse events) | 12 months
  Safety will be measured by careful and comparative evaluation of adverse effects in both groups.
Recurrent biliary obstruction (RBO) | 12 months
  Recurrent biliary obstruction (RBO) has been defined as a composite endpoint of either occlusion or migration.

SECONDARY OUTCOMES:
Clinical success | 2 weeks
  Resolution of jaundice or drop in total bilirubin level by > 50% within 2 weeks after the EUS-CD.
Technical success | 24 hours.
  Technical success was defined as successful placement of the LAMS between the bile duct and the duodenal lumen, creating a transmural ostomy. To evaluate the correct position of the transmural stent, the deployment of the internal flap in the lumen of the bile duct must be verified by ultrasound vision and the internal flap by endoscopic vision.
Survival | 12 months
  Survival is defined as the time elapsed between biliary drainage and the end of follow-up, either due to death and cessation of follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderloni A, Fugazza A, Troncone E, Auriemma F, Carrara S, Semeraro R, Maselli R, Di Leo M, D'Amico F, Sethi A, Repici A. Single-stage EUS-guided choledochoduodenostomy using a lumen-apposing metal stent for malignant distal biliary obstruction. Gastrointest Endosc. 2019 Jan;89(1):69-76. doi: 10.1016/j.gie.2018.08.047. Epub 2018 Sep 4. PMID 30189198
- [Result] El Chafic AH, Shah JN, Hamerski C, Binmoeller KF, Irani S, James TW, Baron TH, Nieto J, Romero RV, Evans JA, Kahaleh M. EUS-Guided Choledochoduodenostomy for Distal Malignant Biliary Obstruction Using Electrocautery-Enhanced Lumen-Apposing Metal Stents: First US, Multicenter Experience. Dig Dis Sci. 2019 Nov;64(11):3321-3327. doi: 10.1007/s10620-019-05688-2. Epub 2019 Jun 7. PMID 31175495
- [Result] Jacques J, Privat J, Pinard F, Fumex F, Chaput U, Valats JC, Cholet F, Jezequel J, Grandval P, Legros R, Lepetit H, Albouys J, Napoleon B. EUS-guided choledochoduodenostomy by use of electrocautery-enhanced lumen-apposing metal stents: a French multicenter study after implementation of the technique (with video). Gastrointest Endosc. 2020 Jul;92(1):134-141. doi: 10.1016/j.gie.2020.01.055. Epub 2020 Feb 19. PMID 32084411
- [Result] Tsuchiya T, Teoh AYB, Itoi T, Yamao K, Hara K, Nakai Y, Isayama H, Kitano M. Long-term outcomes of EUS-guided choledochoduodenostomy using a lumen-apposing metal stent for malignant distal biliary obstruction: a prospective multicenter study. Gastrointest Endosc. 2018 Apr;87(4):1138-1146. doi: 10.1016/j.gie.2017.08.017. Epub 2017 Aug 24. PMID 28843583
- [Derived] Sumalla-Garcia A, Aparicio-Tormo JR, Pedraza-Sanz R, Sanchiz-Soler V, De-la-Serna Higuera C, Andujar X, Vazquez-Sequeiros E, Puigcerver-Mas M, Martinez-Moreno B, Barbera T, Capilla-Lozano M, Martinez-Ortega A, Foruny-Olcina JR, Luna-Rodriguez D, Garcia-Lerma E, Penafiel J, Busquets Barenys J, Laquente-Saez B, Perez-Miranda M, Videla S, Loras C, Gornals JB; Spanish Working Group on Endoscopic Ultrasound Biliary Drainage. Lumen-Apposing Stents With or Without Pigtail in Endosonography-Guided Biliary Drainage for Malignant Distal Biliary Obstruction. Clin Gastroenterol Hepatol. 2025 Jul 21:S1542-3565(25)00611-1. doi: 10.1016/j.cgh.2025.05.025. Online ahead of print. PMID 40701486
- [Derived] Garcia-Sumalla A, Loras C, Sanchiz V, Sanz RP, Vazquez-Sequeiros E, Aparicio JR, de la Serna-Higuera C, Luna-Rodriguez D, Andujar X, Capilla M, Barbera T, Foruny-Olcina JR, Martinez B, Dura M, Salord S, Laquente B, Tebe C, Videla S, Perez-Miranda M, Gornals JB; Spanish Working Group on Endoscopic Ultrasound Guided Biliary Drainage. Multicenter study of lumen-apposing metal stents with or without pigtail in endoscopic ultrasound-guided biliary drainage for malignant obstruction-BAMPI TRIAL: an open-label, randomized controlled trial protocol. Trials. 2022 Feb 25;23(1):181. doi: 10.1186/s13063-022-06106-1. Erratum In: Trials. 2022 Mar 14;23(1):214. doi: 10.1186/s13063-022-06138-7. PMID 35216619